CLINICAL TRIAL: NCT06471569
Title: The Role of Aging and Individual Variation in Exercise Training Responsiveness
Brief Title: Role of Aging and Individual Variation in Exercise Training Responsiveness
Acronym: STRRIDE IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00115833; 5P30AG028716-18 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Prediabetic State; Cardiovascular Diseases; Insulin Resistance; Obesity
Keywords: Exercise; Cardiorespiratory Fitness; Functional Capacity; Cardiometabolic Risk; Physical Reserve; Physical Resilience
MeSH Terms: conditions — Prediabetic State; Cardiovascular Diseases; Insulin Resistance; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Amount/Moderate Intensity (Low/Mod) (Experimental): Six months of low amount/moderate intensity aerobic exercise
  Interventions: Behavioral: Low/Mod
- High Amount/Moderate Intensity (High/Mod) (Experimental): Six months of high amount/moderate intensity aerobic exercise
  Interventions: Behavioral: High/Mod
- High Amount/Vigorous Intensity (High/Vig) (Experimental): Six months of high amount/vigorous intensity aerobic exercise
  Interventions: Behavioral: High/Vig

INTERVENTIONS:
Behavioral: Low/Mod — Aerobic exercise at 50% peak oxygen consumption for the number of weekly minutes prescribed in the original STRRIDE trial
  Arms: Low Amount/Moderate Intensity (Low/Mod)
Behavioral: High/Mod — Aerobic exercise at 50% peak oxygen consumption for the number of weekly minutes prescribed in the original STRRIDE trial
  Arms: High Amount/Moderate Intensity (High/Mod)
Behavioral: High/Vig — Aerobic exercise at 75% peak oxygen consumption for the number of weekly minutes prescribed in the original STRRIDE trial
  Arms: High Amount/Vigorous Intensity (High/Vig)

SUMMARY:
The primary purpose of this study is to assess the effects of aging on markers of physical reserve and exercise-induced adaptations in resilience in older adults who completed a structured exercise program within the last 15 years (Parent trial: STRRIDE-PD; NCT00962962). This feasibility pilot study will enroll up to 26 participants to complete a 6-month aerobic exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who completed participation in the STRRIDE-PD trial (NCT00962962)
* Body Mass Index (BMI) > 18 and < 45 kg/m2
* Stable dose (≥1 month) of any cardiometabolic medications

Exclusion Criteria:

* Poor vein access
* Current use of tobacco or any nicotine products, including e-cigarettes
* Insulin-dependent diabetes
* Active untreated hypothyroidism with thyroid stimulating hormone (TSH) concentrations > 10.0 uIU/mL
* Systemic inflammatory or connective tissue disease, chronic infectious disease, chronic pulmonary disease or symptomatic cardiovascular disease with positive functional study by ECG or imaging
* Current, actively treated malignancy other than dermatologic conditions
* Absolute contraindications to exercise testing: ongoing unstable angina; uncontrolled cardiac arrhythmia with hemodynamic compromise; active endocarditis; symptomatic severe aortic stenosis; decompensated heart failure; acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis; acute myocarditis or pericarditis; acute aortic dissection; physical disability that precludes safe and adequate testing
* Relative contraindications to exercise testing: known obstructive left main coronary artery stenosis; moderate to severe aortic stenosis with uncertain relation to symptoms; tachyarrhythmias with uncontrolled ventricular rates; acquired advanced or complete heart block; hypertrophic obstructive cardiomyopathy with severe resting gradient; recent stroke or transient ischemic attack; mental impairment with limited ability to cooperate; uncorrected medical conditions, such as hypertension, significant anemia, important electrolyte imbalance, and hyperthyroidism
* Modified testing contraindications: acute myocardial infarction (MI) within six months; resting hypertension with systolic or diastolic blood pressures >160/90 mmHg
* Unable to safely participate in an exercise program per study protocol per PI discretion
* Planned, intentional weight loss during study

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | Baseline and post-intervention (~24 weeks)
  Insulin sensitivity will be measured with a 2-hour oral glucose tolerance test
Cardiorespiratory Fitness | Baseline and post-intervention (~24 weeks)
  Cardiorespiratory fitness will be measured with a maximal cardiopulmonary exercise test

SECONDARY OUTCOMES:
Perceived Global Health | Baseline, mid-intervention (~12 weeks), and post-intervention (~24 weeks)
  Self-reported global health will be captured using the Patient-Reported Outcomes Measurement Information System (PROMIS). The questionnaire will be scored using "response pattern scoring" according to the PROMIS scoring manual in order to calculate the T-score for this outcome measure. The population mean T-score for global health is 50, with a score of 40 considered below average and a score of 60 considered above average.
Health-Related Quality of Life | Baseline, mid-intervention (~12 weeks), and post-intervention (~24 weeks)
  Health-related quality of life will be captured using the SF-36 Health Survey. The survey is scored into eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Raw scores will be converted into scale scores ranging from 0 to 100, with higher scores representing better health-related quality of life.
Metabolic Syndrome Z-Score | Baseline, mid-intervention (~12 weeks), and post-intervention (~24 weeks)
  The metabolic syndrome z-score (MSSc) is a continuous weighted score of the five metabolic syndrome variables-fasting high-density lipoprotein cholesterol, triglycerides, glucose, waist circumference, and mean arterial blood pressure. A modified z-score will be calculated for each participant using continuous differences between the Adult Treatment Panel (ATP) III guideline values and participant values with normalization to the cohort's standard deviations. To account for variations in ATP III criteria between men and women, the investigators will use sex-specific MSSc equations. A lower MSSc indicates a better outcome.
Body Composition | Baseline and post-intervention (~24 weeks)
  Body composition will be assessed as percent fat mass and percent fat-free mass.

CONTACTS AND LOCATIONS:
Overall Officials: Leanna M Ross, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No